CLINICAL TRIAL: NCT00229398
Title: Medical and Psychiatric Co-Morbidity Among Treatment Resistant Patients With Major Depression Disorder
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Other Study IDs: SHEBA-99-1744-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Assessing psychiatric and physiological co-morbidity in TRD and non-TRD patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD
* Received at least one adequate treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University